CLINICAL TRIAL: NCT06374602
Title: Efficacy of Pembrolizumab and Lenvatinib in Patients With Anaplastic Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Ernest Dzhelialov, Principal Investigator, Saint Petersburg State University, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33
Record Dates: First submitted 2024-03-27; First posted 2024-04-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Anaplastic Thyroid Cancer
Keywords: Anaplastic thyroid cancer; Immunotherapy; Targeted therapy; Lenvatinib; Pembrolizumab
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Treatment-naive patients with BRAF-negative anaplastic thyroid cancer and previously treated patients, including patients with BRAF-positive anaplastic thyroid cancer (resistant to anti-BRAF therapy).
  Interventions: Drug: Pembrolizumab + Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab + Lenvatinib — Pembrolizumab is a programmed death receptor-1 (PD-1)-blocking antibody. Lenvatinib is Lenvatinib is a kinase inhibitor that inhibits the kinase activities of vascular endothelial growth factor (VEGF) receptors VEGFR1 (FLT1), VEGFR2 (KDR), and VEGFR3 (FLT4).

SUMMARY:
This pilot phase 2 study evaluate the effectiveness and safety of pembrolizumab and lenvatinib in patients with anaplastic thyroid cancer. Patients with anaplastic thyroid cancer who are treatment-naive (BRAF-negative) and who were previously treated with chemptherapy or targeted therapy are scheduled to undergo pembrolizumab and lenvatinib and evaluate the outcomes according to the primary and secondary endpoints.

DETAILED DESCRIPTION:
The aim of the study was to demonstrate the efficacy and safety of pembrolizumab and lenvatinib in patients with anaplastic thyroid cancer.

Scientific hypothesis: the combination of pembrolizumab and lenvatinib is effective and safe in patients with anaplastic thyroid cancer.

Trial design, materials and methods: this study is a pilot Phase 2 study. This study is prospective and open-label. Patients who meet the criteria will be treated with a combination of pembrolizumab and lenvatinib and outcomes will be assessed according to primary and secondary endpoints.

All patients will receive one regimen of antitumor treatment (exploratory therapy). The control will be carried out by monitoring the initial state in dynamics.

Before starting research therapy, data will be recorded for each patient in an individual registration card.

Before starting research therapy, clinical and laboratory parameters will be evaluated and computed tomography of the brain, neck, thoracic and abdominal cavities with intravenous contrast will be performed (initial assessment of the prevalence of the tumor process).

Mutations in the BRAF V600 gene, microsatellite instability (MSI) and PD-L1 expression will be determined in the tumor material (first of all), and the following molecular genetic variants will be determined in the second place (planned): RET, NTRK, ALK, ROS1.

Research therapy includes pembrolizumab 200 mg intravenously for 30 minutes (cycle 21 days) in combination with targeted therapy with lenvatinib 20 mg (2 capsules of 10 mg 1 time per day daily). Dose modification in case of toxicity for pembrolizumab is not provided. For lenvatinib, a sequential dose reduction is provided depending on the previous level (14 mg, 10 mg, 8 mg). When the dose is reduced, a return to the previous level is not carried out.

Duration of treatment: pembrolizumab - up to 35 cycles, until progression or intolerable toxicity, depending on what comes first. Lenvatinib - before progression or intolerable toxicity.

Follow-up period of patients:

follow-up during active treatment within the framework of the study - before progression or intolerable toxicity; patient survival monitoring - documenting subsequent lines of antitumor treatment before the patient's death or loss of contact with him; patient safety monitoring - 30 and 90 days from the date of the final dose.

Assessment of the response to treatment (assessment of clinical and laboratory parameters, computed tomography of the brain, neck, thoracic and abdominal cavities with intravenous contrast) will be carried out monthly or according to clinical indications in the first 6 months, then - according to the decision of the research team. Based on the results of the control study, the response to treatment will be evaluated according to the iRECIST criteria. Patients who meet the criteria for progression will be excluded from the study.

When converting a tumor to resectability and planning surgical treatment, it is recommended to suspend taking lenvatinib at least a week before surgery and resume taking it at least 2 weeks after. There is no relationship between pembrolizumab and complications associated with surgical treatment, and no interruptions in treatment are required.

ELIGIBILITY:
Inclusion Criteria:

* immunohistochemically verified anaplastic thyroid cancer that is not eligible to R0-R1 surgery;
* age ≥ 18 years;
* functional status of ECOG 0-2;
* adequate function of internal organs and bone marrow;
* the ability to give written informed consent.

Exclusion Criteria:

* patients with a mutation in the BRAF V600 gene without previous targeted therapy with BRAF/MEK inhibitors;
* patients with clinically significant hemoptysis and bleeding (for example, from the gastrointestinal tract or tumor-associated bleeding);
* tumor invasion into large vessels;
* patients with open wounds and fistulas;
* contraindications to taking any of the studied drugs;
* patients with poor functional status (ECOG 3-4);
* continuous use of immunosuppressive therapy;
* prior therapy with investigational drugs;
* pregnancy, breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Each month from date of treatment initiation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  The proportion of participants with a partial or complete response to the therapy. It is determined according to the iRECIST criteria.
Progression-Free Survival | 6-month, 1-year, 2-year
  The time from the date of treatment initiation to the radiological progression or death of the patient for any reason.
Safety and Tolerability assessment (Incidence of Treatment-Emergent Adverse Events) | Each visit (every 21 days) assessed up to 48 months
  Safety assessment will be assessed on the basis of adverse events (according to CTCAE 5.0)

SECONDARY OUTCOMES:
Overall survival | 6-month, 1-year, 2-year
  The time from the start date of treatment to the death of the patient for any reason.
The assessment of conversion to resectability | Each month from date of treatment initiation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  The proportion of participants with an initially unresectable or potentially resectable tumor who have moved to a resectable during treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code